CLINICAL TRIAL: NCT06951763
Title: Effect of Myofascial Release on Menstrual Pain Post Caesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan samir Ibrahim, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005675
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stretching exercise group (Active Comparator): The participants will receive stretching exercise program, 3 days/week for 4 weeks.
  Interventions: Other: stretching exrcise
- stretching exercise and myofascial release group (Experimental): The participants will receive same stretching exercises program in addition to myofascial release of cesarean scar, for 30 minutes session twice a week for two weeks.
  Interventions: Other: stretching exrcise; Other: myofascial release

INTERVENTIONS:
Other: stretching exrcise — The participants will receive stretching exercises program for 45 minutes, 3 days/week for 4 weeks.
Other: myofascial release — The participants will receive the same stretching exercises program in addition to myofascial release of cesarean scar, abdominal fascia, diaphragm and psoas muscle for 30 minutes session twice a week for two weeks.
  Arms: stretching exercise and myofascial release group

SUMMARY:
The purpose of this study is to investigate the effect of myofascial release on menstrual pain post cesarean section.

DETAILED DESCRIPTION:
Egypt has the highest cesarean section (CS) rate that has increased from 20% in 2005 to 52% in 2014. This exceptionally high CS rate without a corresponding improvement in maternal and child mortality suggests that although CS is available for populations at risk, numbers of medical unjustified CSs are on the rise.

The CS scar is assumed to be related to adverse clinical gynecological symptoms such as intermenstrual bleeding, dysmenorrhea, dyspareunia and chronic pelvic pain.The incidence of postpartum dysmenorrhea was significantly higher in the cesarean section delivery than in the vaginal delivery.

Cesarean scars have direct links to the perineal fascia and its connection with the transversalis fascia. These scars can interfere with fascial load distribution, which create adhesions to neighboring tissues, the abdominal and pelvic viscera and surrounding anatomical structures are then potentially disrupted, causing inadequate nutrition and inappropriately distributed tension among the various structures affected.

Fascial restrictions obviously decrease blood flow by vascular compression. When the dermis and fasciae are affected by a scar, the sliding structure of the fasciae is altered and when the scar tissues are not capable of adapting to the new stressor, their function is impaired.

MFR procedure lead to vasodilation by increasing capillary permeability. MFR directs force to fascial fibroblasts, as well as indirect strains applied to nerves, blood vessels, the lymphatic system and muscles. There is lacking of studies at this point, so the aim of the study is to investigate the effect of myofascial release on menstrual pain post CS.

ELIGIBILITY:
Inclusion Criteria:

* Women complaining of menstrual pain post - caesarean section (CS).
* Their age will range from 20 to 35 years.
* Their body mass index will range from 20-30 kg/m2.
* Women who gave birth once or twice.
* Women who had C-section 6 weeks to 6 months ago.

Exclusion Criteria:

* Active infection/ infectious skin disease, burn or scars.
* Less than six weeks after CS.
* Any abdominal surgeries other than CS.
* Any spinal deformity as scoliosis or kyphosis.
* History of cancer or radiation to the abdominopelvic region.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Menstrual pain intensity measurement | 4 weeks
  The pain level of each subject will be assessed during menstruation before participation and after the end of the procedure using the visual analogue scale (VAS) by marker across 100 mm line, Participants were asked to put a mark on the line that they felt represented the most severe pain that experienced during menstruation. The following cut points on the pain VAS will be done: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
Menstruation aspects assessment | 4 weeks
  Assessment will be done by WaLIDD questionnaire that included 1) number of anatomical pain locations, 2) Wong-Baker pain range, 3) number of days of pain during menstruation, 4) frequency of disabling pain to perform their activities, e Each tool's variable provided a specific score between 0 and 3, and the final score ranged from 0 to 12 points (Score: 0 without dysmenorrhea, 1-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 severe dysmenorrhea.
Abdominal tenderness assessment | 4 weeks
  Assessment of abdominal tenderness will be done by using the pressure algometer on day 1 and day 3 of menstruation. A one cm2 pressure probe will be positioned perpendicularly to the skin and pressed at a rate of 30kPa/s on specific PPT marked point on the abdomen around the umbilical scar and lumbar region as follows: Two measurements 4cm from the umbilicus, bilaterally (points I and II), two other measurements 4cm below the previous ones (points III and IV), a single measurement 4cm from the lower margin of the umbilicus (point V) and another single measurement into the medial side of the lumbar region below the fifth lumbar vertebra, corresponding to S2-S4 (point VI).
  Participants will be instructed to say "now" when they first felt pain due to the increased pressure. At this point, the algometer will immediately stop and automatically record the amount of pressure applied. Two measures will be collected for each area, with 30s between points testing

SECONDARY OUTCOMES:
Scar tissue mobility assessment: | 4 weeks
  The adherometer will be used to measure scar mobility before and after the procedure for each woman in both groups. An adherometer is a clear plastic sheet with concentric circles, with good reliability on measuring tissue mobility of C-section scars in superior, inferior, left and right directions. Participants will lay supine on a plinth with arms at their sides and legs straight. Marks will be made on the CS scar at 2.5 centimeter (cm) intervals using ruler. The examiner will use the marks to measure tissue extensibility in millimeters (mm) in all four directions.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Kamel, Professor, Study Director — Al-Azhar University; Doaa Osman, As professor, Study Chair — Cairo University
Locations (1):
- Nourhan Samir Ibrahim, Cairo, Egypt